CLINICAL TRIAL: NCT02747329
Title: A Prospective, Multicenter, Randomized Comparative Evaluation of BuMA Supreme Stent and of Xience Stent in Terms of the Extent of Neointimal Formation at 1 Month and 2 Months Via OCT After Implantation in High Bleeding Risk CAD Patients（PIONEER-II OCT Study）
Brief Title: A Comparative Evaluation of the Extent of Neointima Formation at 1 Month and 2 Months After Implantation Using OCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIONEER-II OCT
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease; Stable Angina Pectoris; Unstable Angina Pectoris
Keywords: BuMA Supreme; Xience V/Prime; OCT; neointima formation; HT Supreme
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Angina, Unstable; Neointima

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1st month OCT group implanted BuMA Supreme™ stent (Experimental): This group contains 20 subjects. All subjects in this group will undergoing implantation of BuMA Supreme™ stent. The Primary Endpoint of this group is 1st month QCA and OCT assessment.
  Interventions: Device: BuMA Supreme™ stent
- 1st month OCT group implanted Xience V/Prime stent (Active Comparator): This group contains 20 subjects. All subjects in this group will undergoing implantation of Xience V/Prime stent. The Primary Endpoint of this group is 1st month QCA and OCT assessment.
  Interventions: Device: Xience V/Prime stent
- 2st month OCT group implanted BuMA Supreme™ stent (Experimental): This group contains 20 subjects. All subjects in this group will undergoing implantation of BuMA Supreme™ stent. The Primary Endpoint of this group is 2st month QCA and OCT assessment.
  Interventions: Device: BuMA Supreme™ stent
- 2st month OCT group implanted Xience V/Prime stent (Active Comparator): This group contains 20 subjects. All subjects in this group will undergoing implantation of Xience V/Prime stent. The Primary Endpoint of this group is 2st month QCA and OCT assessment.
  Interventions: Device: Xience V/Prime stent

INTERVENTIONS:
Device: BuMA Supreme™ stent
  Arms: 1st month OCT group implanted BuMA Supreme™ stent; 2st month OCT group implanted BuMA Supreme™ stent
Device: Xience V/Prime stent
  Arms: 1st month OCT group implanted Xience V/Prime stent; 2st month OCT group implanted Xience V/Prime stent

SUMMARY:
The objective of this study is a comparative evaluation of BuMA Supreme™ stent and of Xience V/Prime stent in terms of the extent of neointima formation at 1 or 2 months after implanting in relatively high bleeding risk patients with coronary artery disease using OCT.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, non-inferiority study, which will enroll a total of 80 subjects from approximately 8 centers. All subjects will be firstly randomly assigned to 1st month OCT (40 pts) or 2nd month OCT group(40 pts). Then both two groups will be randomly assigned to undergoing implantation of BuMA Supreme™ stent (20 pts) or Xience V/Prime stent (20 pts). If non-inferiority was met, superiority test will be planned.

All of the patients be followed up to 2 years. The follow-up visits will be conducted at 1 or 2 months (including QCA/OCT investigation), 3 months, 6 months, 1 and 2 years post percutaneous coronary intervention(PCI),in order to observe the Primary Endpoint and Secondary Endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 85 years.
2. Evidence of myocardial ischemia without raised troponin (e.g. stable or unstable angina, silent ischemia demonstrated by positive territorial functional study).
3. Any one or more situation listed below can be considered the patient at high bleeding risk by the doctor:

   * Adjunctive oral anticoagulation treatment planned to continue after PCI；
   * Baseline Hb ≥11 g/dl (or anemia requiring TF during the prior 4 weeks)；
   * Any prior intra-cerebral bleed at any time；
   * Any stroke during the past year；
   * Hospital admission for bleeding during the prior 12 months；
   * Non-skin cancer diagnosed or treated ≤ 3 years；
   * Planned daily NSAID (other than aspirin) or steroids for ≥ 30 days after PCI；
   * Planned major surgery (within 1 year)；
   * Renal failure (calculated creatinine clearance ≥ 40 ml/min)；
   * Thrombocytopenia (≥ 100,000/mm3)；
   * Severe chronic liver disease (variceal hemorrhage, ascites, hepatic encephalopathy or jaundice)；
   * Expected non-compliance to prolonged DAPT for other medical (nonfinancial)reasons ；

     * NSAID, Non-steroidal anti-inflammatory drug; TF, blood transfusion.
4. The patient has a planned intervention of up to two de novo lesions, in different epicardial vessels.
5. Lesion(s) must have a visually estimated diameter stenosis of ≥70% and <100%.
6. Reference Vessel Diameter (RVD) must be between 2.5- 4.0mm, and the vessel length must be no more than 40 mm.
7. Written informed consent.
8. The patient and the patient's physician agree to the follow-up visits including angiographic follow-up and OCT controls at 1 or 2 month.

Exclusion Criteria:

1. Evidence of ongoing acute myocardial infarction in ECG prior to procedure.
2. Left ventricular ejection fraction (LVEF) <30%.
3. The patient is a recipient of a heart transplant.
4. Known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, antiplatelet medication specified for use in the study (clopidogrel and ticlopidine), sirolimus or stainless steel, cobalt metal or sensitivity to contrast media, which cannot be adequately pre-medicated.
5. Other medical illness (e.g. skin cancer diagnosed or treated > 3 years, neurological deficiency) or known history of substance abuse (alcohol etc.) as per physician judgment that may cause non-compliance with the protocol or confound the data interpretation or is associated with a limited life expectancy.
6. Pregnant or breastfeeding woman or woman in fertile period not taking adequate contraceptives
7. Chronic total occlusion(TIMI 0), left main lesion, intervention-required three-vessel lesions, branch vessel diameter ≥ 2.5mm and bypass lesion
8. Patients expected not to comply with 1 month DAPT；
9. Compliance with long-term single anti-platelet therapy unlikely；
10. Active bleeding at the time of inclusion；
11. Patients requiring a planned staged PCI procedure more than one week after theindex procedure；
12. Procedure planned to require non-study stents, or stand alone POBA or stand-alone atherectomy；
13. Reference vessel diameter <2.25 - >4.0mm, vessel length >40mm；
14. Cardiogenic shock；
15. Participation in another clinical trial (12 months after index procedure).
16. Those who is not suitable to attend this trial after the evaluation by the doctor.

OCT exclusion criteria

* Severe tortuous, calcified or angulated coronary anatomy of the study vessel that in the opinion of the investigator would result in suboptimal imaging or excessive risk of complication from placement of an OCT catheter
* Total occlusion or thrombolysis in myocardial infarction(TIMI) flow 0, prior to wire crossing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
The percentage of the struts' neointimal coverage (%) at 1 or 2 months follow-up by OCT assessment. | 1 or 2 months
  1 month OCT assessment is suitable for 1st month OCT group and 2 months OCT assessment is suitable for 2nd month OCT group

SECONDARY OUTCOMES:
Neointimal hyperplasia area/volume | 1 or 2 months
  1 month OCT assessment is suitable for 1st month OCT group and 2 months OCT assessment is suitable for 2nd month OCT group
Mean/Minimal Stent diameter/area/volume | 1 or 2 months
  1 month OCT assessment is suitable for 1st month OCT group and 2 months OCT assessment is suitable for 2nd month OCT group
Mean/Minimal Lumen diameter/area/volume | 1 or 2 months
  1 month OCT assessment is suitable for 1st month OCT group and 2 months OCT assessment is suitable for 2nd month OCT group
Mean/maximal thickness of the struts coverage | 1 or 2 months
  1 month OCT assessment is suitable for 1st month OCT group and 2 months OCT assessment is suitable for 2nd month OCT group
Incomplete strut apposition | 1 or 2 months
  1 month OCT assessment is suitable for 1st month OCT group and 2 months OCT assessment is suitable for 2nd month OCT group
Minimal Lumen Diameter(MLD) and Diameter stenosis percentage(%DS) post procedure and at 3 months | 1 or 2 months
  1 month OCT assessment is suitable for 1st month OCT group and 2 months OCT assessment is suitable for 2nd month OCT group
Late Lumen Loss | 1 or 2 month
  1 month OCT assessment is suitable for 1st month OCT group and 2 months OCT assessment is suitable for 2nd month OCT group
Binary Restenosis (DS ≥50%) | 1 or 2 months
  All measurements will be made of the in-stent, in-segment, proximal and distal stent margins.
Acute success rate | up to 7 days
  It includes the device success,lesion success and procedural success.
Device-oriented Composite Endpoints and its individual components | 1 or 2, 3, 6 months, 1 year, 2 years
  Device-oriented Composite Endpoint (DoCE) is defined as cardiac death, Myocardial Infarction(MI) not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization.
Stent thrombosis according to the ARC definitions | 1 or 2, 3, 6 months, 1 year, 2 years
  Definite and probable stent thrombosis during acute, subacute, later and very late phase.
bleeding events | 1 or 2, 3, 6 months, 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Y Chen, Ph.D., Principal Investigator — the PLA General Hospital
Locations (1):
- The PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li B, Jin QH, Chen YD, Wang CQ, Shi B, Su X, Fu GS, Wu YQ, Zhou XC, Yuan ZY. A prospective, multicenter, randomized OCT study of early neointimal condition at first and second months after BuMA Supreme stent versus XIENCE stent implantation in high-bleeding-risk coronary artery disease patients: study protocol for a randomized controlled trial. Trials. 2019 Jun 7;20(1):335. doi: 10.1186/s13063-019-3361-0. PMID 31174600